CLINICAL TRIAL: NCT05340803
Title: Sedation of Ventilated Traumatic Brain Injury Patients With Midazolam Alone Versus Combination With Dexmedetomidine or Magnesium Sulfate; Monitored by Ultrasonograghic Optic Nerve Sheath Diameter
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alshymaa Hassan Mohammed, Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ONSD for TBI patients
Record Dates: First submitted 2022-04-17; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: TBI (Traumatic Brain Injury)
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Midazolam; Dexmedetomidine; Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: To compare use of midazolam alone versus combination of midazolam with dexmedetomidine or magnesium sulfate in patients with sever TBI ( Glasgow Coma Scale < 8 and in need for mechanical ventilation) as regards effect on ICP monitored by US-ONSD as the primary outcome and anti-inflammatory effect (neuroprotective effect) by measurement of serum IL-6 as a secondary outcome.
Who Masked: Participant, Outcomes Assessor
Masking Description: Each group will contain 36 patients by double-blind manner using numbered sealed envelopes and the main investigator responsible for measurement ONSD will not be informed about the drug or drugs used for each patient
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): Sedation by midazolam alone
  Interventions: Radiation: Ultrasonograghic optic nerve sheath diameter US-ONSD; Drug: midazolam
- Group B (Active Comparator): Sedation by midazolam and dexmedetomidine during the first 24 hours
  Interventions: Radiation: Ultrasonograghic optic nerve sheath diameter US-ONSD; Drug: midazolam; Drug: dexmedetomidine
- Group C (Active Comparator): Sedation by midazolam and magnesium sulfate during the first 24 hours
  Interventions: Radiation: Ultrasonograghic optic nerve sheath diameter US-ONSD; Drug: midazolam; Drug: magnesium sulfate

INTERVENTIONS:
Radiation: Ultrasonograghic optic nerve sheath diameter US-ONSD — To compare effect of sedation in 3 groups by follow up of intracranial pressure by US-ONSD
Drug: midazolam — midazolam
Drug: dexmedetomidine — dexmedetomidine
  Arms: Group B
Drug: magnesium sulfate — magnesium sulfate
  Arms: Group C

SUMMARY:
In TBI, there is a strong correlation between increased ICP and bad outcome. So, appropriate monitoring can be the gold standard in management of TBI. ICP can be measured by invasive and noninvasive methds. One of these noninvasive methods is bedside measurement of optic nerve sheath diameter (ONSD) by ocular ultrasonography

DETAILED DESCRIPTION:
In the previous few years, agreat evidence has established for efficiency of dexmedetomidine (DEX) in management of TBI. Dexmedetomidine is a highly selective alpha-2 receptor agonist, its major sympatholytic and sedative actions are mediated primarily via reduced transmission in the locus coeruleus which is a part of the reticular activating system. It provides excellent sedation without respiratory depression, ease of arousability, and need not be stopped during weaning the patient from mechanical ventilation or for neurological assessment. It suits as an ideal sedative agent for patients with TBI. DEX has been shown to reduce cerebral ischemia/ reperfusion injury by suppressing inflammation, activating the anti-apoptotic signaling pathways, and inhibiting neuronal autophagy. Animal studies have shown that alpha-2 agonists are neuroprotective in craniocerebral and subarachnoid injuries but this has not been definitively shown in humans . The efficacy of DEX for sedation in intubated ICU patients is well established; however, its use in patients with TBI has not been comprehensively described .

Magnesium has shown great promise as a potential therapeutic agent in TBI during animal experiments . Magnesium is essential for the maintenance of cell membrane integrity, the stabilisation of genetic material and for a number of fundamental enzymatic reactions such as glycolysis, oxidative phosphorylation and protein synthesis, it is also known to act presynaptically to inhibit the release of excitatory amino acids, and be a non-competitive inhibitor of the voltage-gated N-methyl-D-aspartate (NMDA) receptor, an important link in the excitotoxic phase of secondary brain injury. As a consequence, magnesium's role in TBI has been of great interest to researchers.

ELIGIBILITY:
Inclusion Criteria:

1. Middle age patients ( 18- 45 years old).
2. Sever TBI (GCS < 8 and in need for mechanical ventilation).
3. Stable hemodynamics

Exclusion Criteria:

1. Age: younger than 18 or older than 45 years old.
2. Mild and moderate TBI (GCS > 8).
3. Shocked and hypoxic patients.
4. Contraindications to dexmedetomidine as sever hypotension (mean arterial blood pressure < 60 mmHg), sever bradycardia (heart rate < 45 beat/min), and AV block in the group that will be sedated by midazolam and dexmedetomidine (group B).
5. Adverse effects of dexmedetomidine in group B and need to stop it as sever hypotension (mean arterial blood pressure < 60 mmHg) , sever bradycardia (heart rate < 45 beat/min), and atrial fibrillation.
6. Contraindications to magnesium sulfate as heart block, myocardial damage, hypermagnesemia and renal failure in the group that will be sedated by midazolam and magnesium sulfate (group C).
7. Manifestations of magensium toxicity in group C and need to stop infusion if urine output < 80 mL in 4 hours, deep tendon reflexes are absent or serum magnesium level > 3.5 mmol/L .

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Optic nerve sheath diameter (ONSD) changes by using ultrasound | up to 24 hours
  ONSD is an indicator for changes in intracranial pressure in response to sedation with midazolam alone versus combination with dexmedetomidine or magnesium sulfate which group will show better control of the increased intracranial pressure to prevent secondary brain insults. ONSD of 5.8mm was used as cutoff point for identifying ICP above 20 mmHg.